CLINICAL TRIAL: NCT02963532
Title: A Direct Comparison of Predictors for Extubation in Children Less Than 7 Years Old Undergoing Anesthesia: A Prospective Observational Study
Brief Title: Extubation in Pediatric Patients: An Observational Study
Status: Completed | Type: Observational
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Other Study IDs: 00039203
Record Dates: First submitted 2016-11-08; First posted 2016-11-15 (Estimated); Last update posted 2018-01-08 (Actual); Status verified 2017-01

CONDITIONS: Anesthesia, Pediatric

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: We are observing criteria present at extubation — We will not be performing any intervention. We will only be observing what clinical data is present at the time of extubation and how predictive are different pieces of clinical data.

SUMMARY:
The timing of extubation following surgery and anesthesia in young children is a complex decision frequently guided by the experience of the clinician. The clinician frequently must make a decision based on assimilating multiple cues that may or may not demonstrate that the patient is ready for extubation such as eye opening, conjugate gaze, spontaneous ventilation, and end tidal agent concentration. At this time there is no published data on the predictive ability of individual extubation criteria for young patients undergoing anesthesia for surgery so most practice is based solely on experience and anecdotal teaching. In some cases if the timing is misjudged and the patient is extubated too early negative airway reflexes such as breath holding and laryngospasm may take over creating a critical situation in which the patient forgoes gas exchange and rapidly desaturates with the potential for bradycardia and further cardiovascular collapse.

Routine criteria used to determine fitness for extubation have been primarily described in the intensive care unit literature and may be less relevant in the operating room in the setting of routine general anesthetics. Most predictors including adequate tidal volume, presence of conjugate gaze, eye opening, patient movement purposeful or otherwise, low end tidal anesthetic agent concentration, response to physical or verbal stimulation and the laryngeal stimulation test have not previously been evaluated to determine their individual predictive value in deciding if the presently anesthetized patient now emerging is ready to be extubated.

In order to perform a laryngeal stimulation test the patient must be breathing spontaneously and practitioner will gently move the endotracheal tube up and down stimulating the larynx. In patients in stage 2 of anesthesia, the clinician will typically observe a cough or series of coughs followed by a respiratory pause of greater than 5 seconds. In this situation the patient has not adequately passed through stage 2 and remains at increased risk for apnea, breath holding, or laryngospasm. If the patient is in stage 1 of anesthesia the clinician will observe a cough followed by a brief pause (less than 5 seconds) or almost immediate return to spontaneous ventilation.

In conclusion, their exist no quantitative data on the predictive value of these various criteria for extubation and the goal of our study is determine the indivdual predictive value of different criteria in determing fitness for extubaion in young pediatric patients by recording the presence or absence of various criteria in pediatric patients at the time of extubation during routine anesthetic care.

DETAILED DESCRIPTION:
Objectives

The objective of this study is to prospectively observe the frequency and predictive value of specific signs and criteria and correlate those with successful extubation in young children to determine which are present with the greatest frequency and which signs are most predictive of successful extubation.

Methods and Measures

Design

A trained observer will prospectively observe emergence and extubation in pediatric patients between the ages of less than 7 years of age in which potent inhalational agents were used for anesthetic maintenance. They will record the presence or absence of certain accepted signs that a young child is ready for extubation such as eye opening, postive larygneal stimulation test, purposeful movement, end tidal agent concentration, and several others (see Appendix 1 for complete list). We will also record the use of nondepolarizing neuromuscular blocking drugs, use and presence of train of four monitoring, and end tidal carbon dioxide concentration at the time of extubation. Timing of extubation will be at the discretion of the attending anesthesiologist caring for the patient according to their usual practice. Following extubation we will observe the patient and a second checklist will be filled out detailing any events such as the need for continuous positive pressure with 100% oxygen, reintubation. The quality of extubation will be scored as either "successful," "moderately successful," or "failed," according to predefined criteria; see appendix 1.The investigators will record the oxygen saturation, respiratory rate, and presence or absence of additional oxygen supplementation such as "blow by," "mask oxygen" or "nasal cannula" on arrival to the Post anesthesia care unit, at 5, 10, and 30 minutes after arrival in the post anesthesia care unit. The investigators will also record the post anesthesia care unit length of stay as defined as the time at arrival until the time the nurse deems that the patient has recovered sufficiently to leave the post anesthesia care unit either for home or for their inhouse bed.

Investigators will record age, height, weight, gender, American society of anesthesiologist status, type of surgery, and presence or absence of any upper respiratory infection symptoms in the previous 2 weeks, and any premedication, type of inhalational agent used.

Investigators will observe patients less than 7 years old based on the operating room schedule.

The study will be performed at Wake Forest Baptist Medical Center a tertiary academic medical center.

Subjects selection criteria

Pediatric patients under the age of 7 scheduled for surgery and anesthesia with an endotracheal tube will be observed at the time of extubation.

• Inclusion Criteria

Patients less than 7 years of age scheduled for surgery and anesthesia in which an endotracheal tube is placed for airway management and potent inhalational agents are used for anesthetic maintenance for which a trained study observer can be present for extubation will be included.

• Exclusion Criteria

Patients using a laryngeal mask airway or other supralaryngeal device for airway management during an elective procedure.

Patients with a tracheostomy in place. Any case in which total intravenous anesthesia is used. Patient in which a mask alone is used for airway management.

• Sample Size

Using an a priori sample size calculator for multiple regression analysis based on effect size f2 of 0.05 in a model with 7 predictors, a probablility level of 0.05, and a statistical power of 80% we estimate a sample size of 293 patients. The calculator can be found at the following internet address: http://www.danielsoper.com/statcalc/calculator.aspx?id=1 Given the number of 293 patients we will observe 300 extubations.

Interventions and Interactions:

Interventions and interactions for the patient should be minimal since this is an observational study. Study personnel will monitor the pediatric operating room schedule during the day to look for cases where an endotracheal tube is being used for airway management in children less than 7 years of age. Study personnel will consult with the responsible anesthesia team and will prospectively record data at the time of emergence and extubation. They will also intermittently observe the patient in the post anesthesia care unit but may delegate the recording of respiratory data in the post anesthesia care unit at arrival, 5, 10, and 30 minutes. They will also record post anesthesia care unit length of stay.

Outcome Measure(s)

Outcome measures will be successful, moderately successful or failed extubation and the correlation, frequency, and predictive value of individual subjective and objective criteria for extubation.

Analytical Plan

Results will be analyzed initially using descriptive statistics and multivariate logistic regression analysis to determine the predictive value of different criteria for successful extubation and further to determine if one criteria is more predictive than another.

Human Subjects Protection

Subject Recruitment Methods

Study participants will be identified by looking at the pediatric operating room schedule and consulting with the anesthesia team responsible for the patient to determine if they used an endotracheal tube for airway management and then further if they plan to extubate the patient at the end of the procedure. If the aforementioned is acceptable and the patient meets the age inclusion criteria and a member of the study is available they will observe the emergence and record data based on what is occurring during the emergence and extubation.

Informed Consent

Informed consent will not be sought as this is an observational study designed to observe criteria used in the routine practice of pediatric anesthesia to determine the timing of extubation. All clinical care will be administered at the discretion of the attending anesthesiologist according to their routine standard practice.

ELIGIBILITY:
Inclusion Criteria:

* Patients less than 7 years of age scheduled for surgery and anesthesia in which an endotracheal tube is placed for airway management and potent inhalational agents are used for anesthetic maintenance for which a trained study observer can be present for extubation will be included.

Exclusion Criteria:

* Patients using an LMA or other supralaryngeal device for airway management during an elective procedure.
* Patients with a tracheostomy in place.
* Any case in which total intravenous anesthesia is used.
* Patient in which a mask alone is used for airway management.

Ages: 1 Month to 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Pediatric Patients < 7 years of age.
Sampling Method: Probability Sample
Enrollment: 600 (Actual)
Dates: Start 2016-12 (Actual); Primary Completion 2017-12-04 (Actual); Study Completion 2017-12-04 (Actual)

PRIMARY OUTCOMES:
Quality of Extubation. Defined as: Successful, Moderately Successful, or Failed. | This will be observed at the time of extubation.
  Successful is defined as oxygen saturation >92% and requires continuous positive airway pressure with 100% oxygen < 1 minute. Moderately successful:continuous positive airway pressure for >1 minute with 100% oxygen, inspiratory stridor without sequelae, oxygen saturation <92% for > than 30 seconds, failed: patient required reintubation, laryngospasm, breath holding > 10 seconds, requires continuous positive airway pressure > 2 minutes with 100% oxygen.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Templeton, MD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No